CLINICAL TRIAL: NCT04073914
Title: Type 1 Teamwork: A Tool for Parents of Adolescents With Type 1 Diabetes
Acronym: Type1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R44DK098857 (NIH)
Record Dates: First submitted 2019-03-11; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-02

CONDITIONS: Type1diabetes; Type1 Diabetes Mellitus
Keywords: Diabetes; Adolescence; Parents
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: To evaluate the complete program the investigators conducted a modest randomized clinical trial, randomizing parents to the Type1Teamwork program or a wait-list control group. Results were analyzed using general linear repeated measures models with training group, and time as fixed effects. The primary hypotheses comparing changes in domain totals over time will be tested by the interaction effect of time by treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Type 1 Teamwork program
  Interventions: Behavioral: Type 1 Teamwork Program
- Control (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Type 1 Teamwork Program — Psychoeducational web program
  Arms: Intervention

SUMMARY:
Type 1 Diabetes (T1DM) is a common chronic illness in children which presents difficult and often stressful management concerns for parents. As children approach adolescence, this burden increases with the desire for independence and self-management. No tool exists that addresses in a user friendly, easy to access and socio-culturally appropriate way, the psychosocial needs of parents as they move through this transition. This program targets the parents to help them at the very point where this transition is occurring.

DETAILED DESCRIPTION:
Type 1 diabetes (T1D) is one of the most common chronic illnesses in children, affecting 1 in 400,1 with evidence that its prevalence is increasing worldwide.2 The prevalence of T1D in adolescents is approximately 70% White, 22% Hispanic, and 8% Black.3-5 Parents of children with T1D are responsible for a labor-intensive and complicated daily regimen that has been described as an overwhelming experience, requiring constant vigilance.6 Intensive management of T1D requires frequent blood glucose monitoring, multiple insulin injections or use of an insulin pump, frequent alterations in insulin dose to match changing diet and activity patterns, and regular visits to health care providers. This 24/7 attention to their child's health manifests in elevated rates of parental perception of stress and increased risk for depression and anxiety. The prevalence of anxiety symptoms for parents of children with T1D range from 21-59%; depressive symptoms from 10-74%; psychological distress from 29-33%; and posttraumatic stress symptoms from 19-24%.7-9 Parental psychological distress has negative health implications for the parent, the overall functioning of the family, the psychological adjustment of their child with T1D, diabetes management, and child metabolic control.10-14 The goal of this application is to complete the psycho-educational web-based program for parents of adolescents with T1D (Type1Teamwork) which will help to: 1) decrease parental perceived stress and distress; 2) promote parental adjustment to the developmental transitions in adolescence; 3) support adolescent autonomy and transfer of diabetes responsibility from parent to adolescent; 4) decrease family conflict; and 5) maintain metabolic control during adolescence. The investigators propose to complete two major Aims in Phase II:

Specific Aim 1: Develop the Type1Teamwork program (for use on computer, tablet, or smart phone) based on the activities completed in Phase I. Six content themes have been identified as important to parents and providers. Feasibility assessment has provided support of these content themes as well as substantive recommendations to ensure content and interactivity is engaging and meets the needs of parents of children with T1D as well as health care providers. The investigators will use an iterative process of development and evaluation, collaborating with our technology team, parent advisors, and clinical consultants to ensure development of a quality product and to submit a peer reviewed manuscript for publication of the results.

Specific Aim 2: Evaluate the Type1Teamwork program through a modest randomized clinical trial. The investigators will determine the effect of the program on parent psychosocial outcomes (stress, depression, and anxiety), adolescent autonomy, parent-adolescent responsibility for T1D management, family conflict, and adolescent metabolic control. Results will be presented at diabetes meetings, published in top tier journals (to provide clinical and scientific evidence of the newly developed program), and widely disseminated per the commercialization and marketing plan.

ELIGIBILITY:
Inclusion Criteria:

* Parent of an adolescent with T1D aged 11-16;
* Able to comply with the terms of the trial (available time commitment);
* Able to speak, read, and write in English

Exclusion Criteria:

• Not meeting inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2018-03-26 (Actual); Study Completion 2018-03-26 (Actual)

PRIMARY OUTCOMES:
Change in Parent Stress using the Perceived Stress Scale (PSS) | Baseline, 3 months, and 6 months
  Participants of the Type1Teamwork program will have a significant decrease in parent stress compared to the control arm participants at 3 and 6 month follow-up. The researchers are using the PSS, a 14-item scale that measures a person's perceived stress by considering the degree to which situations in one's life are appraised as stressful. Items evaluate how unpredictable, uncontrollable, and overloaded respondents find their lives. Higher scores indicate greater perceived stress. Chronbach's alpha was 0.89 in our sample. REF: Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. Journal of health and social behavior. Dec 1983;24(4):385-396.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Marceau, MPH, Principal Investigator — Carelon Research
Locations (2):
- United States (2):
  - Yale University, New Haven, Connecticut
  - New England Research Institutes, Watertown, Massachusetts

IPD SHARING:
Plan to Share IPD: No